CLINICAL TRIAL: NCT02738658
Title: Comparison of the Vasomotor Function and Myocardial Flow in Patients Treated
Brief Title: Comparison of the Vasomotor Function and Myocardial Flow in Patients Treated With Bioresorbable and Metallic Stents at 1 Year
Acronym: BVS-Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Josep Gomez Lara, MD, PhD, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20151810
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Stable Angina
Keywords: Coronary microcirculatory dysfunction; Coronary endothelium dysfunction
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioresorbable vascular scaffold (BVS) (Experimental): Patients with stable coronary angina with coronary artery disease suitable to be treated with a bioresorbable vascular scaffold.
  Interventions: Device: Bioresorbable vascular scaffold
- Everolimus-eluting stent (EES) (Active Comparator): Patients with stable coronary angina with coronary artery disease suitable to be treated with a Everolimus-eluting stent .
  Interventions: Device: Everolimus-eluting stent

INTERVENTIONS:
Device: Bioresorbable vascular scaffold
  Other Names: Bioresorbable stents
  Arms: Bioresorbable vascular scaffold (BVS)
Device: Everolimus-eluting stent
  Arms: Everolimus-eluting stent (EES)

SUMMARY:
Background: A total of 25-50% of patients with stable coronary atherosclerosis treated with metallic stent implantation remain with effort angina despite optimal medical treatment and absence of stent restenosis at 1 year. The most plausible cause of persistent effort angina after stent implantation is microcirculatory dysfunction. Coronary circulation matches the myocardial blood supply and oxygen consumption. Metallic stent implantation has been related with endothelial dysfunction and impaired coronary blood flow reserve (relation between coronary blood flow at rest and maximal hyperemia) of the treated vessel at 1 year.

Bioresorbable Vascular Scaffold (BVS) has been shown to improve the endothelial function and to improve the angina symptoms at 1 year. However, the coronary blood flow of BVS has never been tested.

Main objective: To determine differences in the blood average peak velocity at maximal hyperemia with adenosine infusion between patients treated with bioresorbable and metallic coronary stents at 1 year after stent implantation.

Methodology: A total of 70 patients are 1:1 randomized to everolimus-eluting metallic stent (EES) versus everolimus-eluting BVS implantation in patients with stable coronary disease. At 1 year, patients undergo to invasive coronary angiography prior cessation of vasomotor drugs. A pressure/Doppler wire is advanced distally to the "treated segment" and the endothelial (acetylcholine) and non-endothelial (adenosine and nitroglycerine) vasomotor function is assessed with quantitative coronary angiography and pressure and Doppler measurements. Angina test questionnaires are obtained at different time-points of the study.

Expected results: A difference between patients treated with BVS and EES of 12.0 cm/sc in the maximal average peak velocity (APV) under maximal hyperemia (with adenosine administration) is expected, as assessed by Doppler measurements, at 1 year after stent implantation. The study is powered to assess superiority in terms of maximal APV favoring patients treated with BVS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina or silent angina with myocardial ischemia detected by non-invasive tests or patients with acute coronary syndromes with no increase of > 5 times the upper value of normality of cardiac biomarkers (troponin).
* Patients with coronary artery disease with angiographic stenosis >

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Difference in the average peak velocity at maximal hyperemia between bioresorbable vascular scaffolds and everolimus-eluting stents as assessed by doppler wire measurement. | 1-year after stent implantation

SECONDARY OUTCOMES:
Difference in endothelial dysfunction with acetyl-choline infusion between bioresorbable vascular scaffolds and everolimus-eluting stents as assessed by quantitative coronary angiography (4% of lumen reduction) | 1-year after stent implantation

OTHER OUTCOMES:
Difference in fractional flow reserve at maximal hyperemia between the two treatment groups as assessed by pressure-wire measurement | 1-year after stent implantation

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinic, Barcelona